CLINICAL TRIAL: NCT00926341
Title: A Study on the Effects of Peroxisome Proliferators Activated Receptor-γ Agonists on Certain Biochemical and Inflammatory Markers in Patients With Metabolic Syndrome
Brief Title: The Effects of Peroxisome Proliferators Activated Receptor-Gamma (PPAR-γ) Agonists on Certain Biochemical and Inflammatory Markers in Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aligarh Muslim University (Other)
Responsible Party: DR.S.F.Haque,Reader,, Department of Medicine, JNMC,AMU
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFH-CASR-FMD-06
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; inflammatory markers; Thiazolidinediones; Angiotensin receptor blockers
MeSH Terms: conditions — Metabolic Syndrome | interventions — Pioglitazone; Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active control (No Intervention): 1. Active Control: (n=20), intervention: no intervention
- PIO arm (Active Comparator): PIO arm (n=30), Pioglitazone 30 mg/day, given for 24 weeks.
  Interventions: Drug: Pioglitazone
- Telmi arm (Active Comparator): Telmia arm (n=30): Tab. Telmisartan 40 mg/day given for 2 weeks.
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Pioglitazone — Tab. Pioglitazone-30 mg/day, oral, 24 weeks
  Arms: PIO arm
Drug: Telmisartan — Tab. Telmisartan- 40 mg/day, oral, 24 weeks
  Arms: Telmi arm

SUMMARY:
Metabolic syndrome, labeled as the world's latest epidemic, is the force behind the global epidemic of Type 2 Diabetes Mellitus and Cardio Vascular Diseases. This emerging epidemic is an important public health problem for South Asians in their homeland and worldwide.

Pharmacological therapy is a critical step in the management of patients with metabolic syndrome. In general, treatment for metabolic syndrome, that targets all or most of the components of metabolic syndrome is either deficient or non-existent. The study presented here is the pioneering work in the management of metabolic syndrome, the emerging global epidemic.

DETAILED DESCRIPTION:
Our understanding of the metabolic syndrome has been improved by the discovery nuclear peroxisome proliferator-activated receptors (PPARs). PPAR-γ is a nuclear receptor that influences the expression of multiples gene involved in carbohydrate and lipid metabolism. At the crossroads of obesity, insulin resistance, and cardiovascular disease is the nuclear receptor PPAR-γ. At present, metabolic syndrome can be described as a 'PPAR-γ agonist resistance syndrome.' The modulation of PPAR-gamma activity is an interesting therapeutic approach to address multi-component metabolic syndrome and its consequent cardiovascular events.

Recent studies have indicated that in addition to anti diabetic properties, PPAR-γ agonists (TZD)-Pioglitazone, provides protection against atherosclerotic cardiovascular disease. Further, the identification of ARBs-Telmisartan and Irbesartan, as capable of activating PPAR - γ, has provided a novel approach in treating hypertension, insulin resistance, hyperlipidemia, and inflammation.

Emerging evidence suggests that PPAR-γ agonist: Thiazolidinediones (TZD)-Pioglitazone is an insulin sensitizer and modulator of metabolic syndrome, through its pleiotropic effects on vascular risk and have beneficial effects on systemic inflammatory markers. Despite the beneficial effects of full PPAR- agonists like the TZDs, recent evidence suggests that full PPAR- agonists are less than optimal agents in patients with metabolic syndrome. TZDs promote adipo-genesis and fluid retention, causing weight gain and precipitate congestive heart failure. The adverse effects of full PPAR- agonists like the TZDs have reinforced the need to identify additional therapies with insulin-sensitizing properties. The recent discovery that telmisartan, an angiotensin II type 1 receptor (AT1-R) blockers (ARBs), is uniquely capable of selective PPAR- -modulating activities, have the potential to treat both hemodynamic and biochemical features of insulin resistance and metabolic Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 3 out of 5 criteria of metabolic syndrome of NCEP-ATP III (Asian-Pacific) guideline:

  1. Waist circumference of > 90 cm in men or > 80 cm in women;
  2. Serum triglycerides of >= 150 mg/dl;
  3. High-density lipoprotein-cholesterol (HDL-C) levels of < 40 mg/dl in men and < 50 mg/dl in women;
  4. Fasting glucose of 6.1/ m.mol (≥l00 mg/dl)
  5. Systolic blood pressure > = 130 mmHg or Diastolic blood pressure >= 85 mmHg or OR on anti-hypertensive therapy
* Ability to perform all tasks related to glycemic control and risk factor management.
* Written informed consent.
* Between 30 and 70 years of age of either sex.

Exclusion Criteria:

* Concomitant use of ACE inhibitor or ARB in the last 3 months. Or angioedema with ACE I / ARB or uncontrolled hypertension (SBP >=160 mmHg and/or DBP >=100 mmHg) or known case of secondary hypertension.
* Patients already taking any thiazolidinediones or having contraindications for the same.
* Class III or IV heart failure
* Renal dysfunction as defined by serum creatinine > 130umol/L (> 2.0 mg/dl)
* Concomitant use of statin or fenofibrate.
* Hepatic dysfunction as defined by SGPT (ALT)> 3 times the upper limit of normal
* Taking Anti-obesity medications/metformin
* History of drug or alcohol dependency within six months.
* History of active malignancy, chronic,inflammatory disorder, or chronic infections which would interfere with protocol completion.
* Use of systemic glucocorticosteroids/aspirin/anti-inflammatory drugs.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Control of blood pressure and decline in triglycerides level | 24 weeks

SECONDARY OUTCOMES:
Improvement in Inflammatory markers Hs-CRP, TNF-alpha, IL-6 and visceral obesity | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shahzad F HAQUE, MBBS.MD, Principal Investigator — Department of medicine,JNMC, AMU, ALIGARH
Locations (1):
- Department of Medicine, J.N.Medical,College, AMU,Aligarh, Aligarh, Uttar Pradesh, India

REFERENCES:
- [Background] Szapary PO, Bloedon LT, Samaha FF, Duffy D, Wolfe ML, Soffer D, Reilly MP, Chittams J, Rader DJ. Effects of pioglitazone on lipoproteins, inflammatory markers, and adipokines in nondiabetic patients with metabolic syndrome. Arterioscler Thromb Vasc Biol. 2006 Jan;26(1):182-8. doi: 10.1161/01.ATV.0000195790.24531.4f. Epub 2005 Nov 10. PMID 16284192
- See also: A Study on the Effect of Peroxisome Proliferators... — http://ahajournals.com